CLINICAL TRIAL: NCT04653025
Title: Immediate Placement and Temporization of Tapered Implants in Extraction Sockets or Early Implant Placement Protocol? A Randomized Controlled Clinical Trial.
Brief Title: Immedaite vs Early Implant Placement in Aesthetic Area
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vilniaus Implantologijos Centro (VIC) Klinika (Network)
Collaborators: Institut Straumann AG (Industry)
Responsible Party: Principal Investigator, Algirdas Puisys, DDS, PhD, Principal investigator, Vilniaus Implantologijos Centro (VIC) Klinika
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIS0816
Record Dates: First submitted 2020-11-19; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Single Implant; Immediate Implant Treatment; Early Implant Treatment

STUDY DESIGN:
Intervention Model Description: Patients with a failing maxillary anterior tooth were included in this study. After atraumatic extraction, test group patients received an immediate implant with provisional restoration, while patients in the control group received an implant after 6 weeks of healing. After 4 months (test group) and 6 months (control group) definitive restorations were delivered. All patients were followed for 1 year post restoration and pink esthetic score (PES), mid-buccal mucosal level (MBML), crestal bone changes (CBC) and peri-implant soft tissue parameters were recorded at several time points. In addition, patient chair time was recorded
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Test group patients received an immediate implant with provisional restoration, bone augmentation and soft tissue grafting
  Interventions: Device: Implant placement
- Control group (Experimental): Patients in the control group received soft tissue grafting after tooth extraction and an implant with bone augmentation after 6 weeks of healing.
  Interventions: Device: Implant placement

INTERVENTIONS:
Device: Implant placement — After tooth extraction implants were placed either immediate or delayed approach

SUMMARY:
The purpose of this randomized clinical trial, of 50 patients in need of a maxillary anterior implant, was to assess the esthetic outcomes of immediate temporization of immediately placed tapered implants in fresh extraction sockets with soft tissue and bone augmentation as compared to early placed implants with conventional loading. Secondary objectives included the influence of immediate provisionalization on the success rate of tapered implants and crestal bone stability.

DETAILED DESCRIPTION:
Patients with a failing maxillary anterior tooth were included in this study. After atraumatic extraction, test group patients received an immediate implant with provisional restoration, while patients in the control group received an implant after 6 weeks of healing. After 4 months (test group) and 6 months (control group) definitive restorations were delivered. All patients were followed for 1 year post restoration and pink esthetic score (PES), mid-buccal mucosal level (MBML), crestal bone changes (CBC) and peri-implant soft tissue parameters were recorded at several time points. In addition, patient chair time was recorded.

ELIGIBILITY:
Inclusion Criteria:

1. no recession of gingival contour of tooth to be extracted,
2. no periodontal bone loss of neighboring anterior teeth,
3. no implants in neighboring teeth,
4. class I extraction socket (intact buccal wall),
5. atraumatic extraction of the tooth with intact socket walls remaining,
6. only one implant per patient to be inserted.

Exclusion Criteria:

1. deep bite (severe II class),
2. systemic disease (diabetes, osteoporosis),
3. heavy smokers (more than 10 cigarettes/day) were excluded.
4. atraumatic extraction of the tooth failed,
5. the primary stability (at least 25 Ncm) needed for implant temporization, after implant placement, was not achieved.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2030-01-10 (Estimated)

PRIMARY OUTCOMES:
Changes of pink aesthetic score (PES) over time | Baseline, 1 year and 5 years after prosthetic delivery
  pink esthetic score means evaluation of seven parameters of anterior tooth aesthetics - mesial and distal papila, soft tissue level, contour, texture, color and convexity. Each parameter may be evaluated by score 0,1 or 2, were the score 0 means the worst outcome, 2 - the best. Evaluation will be performed visually using digital photos.

SECONDARY OUTCOMES:
Changes of marginal bone level (MBL) around implant neck | Baseline, 1 year and 5 years after prosthetic delivery
  Periapical x-rays will be used to measure crestal bone sability distally and mesially of dental implant using certificated x-ray program after calibration. Measurement will be recorded in millimetres from implant neck to the first bone to implant contact
Recession changes of gingiva of restored tooth on the implant | Baseline, 1 year and 5 years after prosthetic delivery
  Mid-buccal recession evaluation will be performed using standardised periodontal probe. Measurement of the crown hight will be done in the middle of the tooth from incisal edge to the highest point and recorded in millimetres.

CONTACTS AND LOCATIONS:
Locations (1):
- VIC clinic, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD